CLINICAL TRIAL: NCT06156137
Title: Characteristics of Blood Glucose Variability in Patients With Type 2 Diabetes Mellitus Complicated With COVID-19 and Its Effect on the Prognosis of the Disease
Brief Title: Characteristics of Blood Glucose Variability in Patients With Type 2 Diabetes Mellitus and COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, kuanxiao Tang, chief physician, Qilu Hospital of Shandong University
Other Study IDs: kuanxiao Tang
Record Dates: First submitted 2023-11-23; First posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: COVID-19 Pneumonia; Type2diabetes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- adverse outcomes: The composite adverse outcomes are defined as either a >20-day length of stay intensive care unit admission, mechanical ventilation use, or death.
  Interventions: Other: Glucose variability
- favorable outcomes: favorable outcomes the patient are defined as discharged with improvement and hospitalization less than 20 days.
  Interventions: Other: Glucose variability

INTERVENTIONS:
Other: Glucose variability — A retrospective cohort study was conducted in hospitalized T2DM patients with NCP who were discharged or died. Clinical data and blood glucose variability parameters were collected by computer blood glucose monitoring technology (CGM). Time in range (TIR), time above target range (TAR), time below target range (TBR), mean amplitude of glycemic excursions (MAGE), absolute mean daily difference (MODD) and other indicators were used.

SUMMARY:
using intermittently scanned continuous glucose monitoring (isCGM) to clarify the characteristics of blood glucose variability parameters in T2DM patients with NCP, guide the formulation of reasonable clinical treatment measures and make timely and reasonable adjustments, improve the prognosis of patients, shorten the length of hospital stay, and reduce medical costs.

The goal of this observational study is to investigate the characteristics of blood glucose variability in patients with type 2 diabetes mellitus (T2DM) complicated with novel coronavirus pneumonia (NCP) and its effect on disease progression and prognosis.

The main question it aims to answer is:After fully lifting coronavirus disease 2019 (COVID-19) pandemic control measures in mainland China in 12/2022, the incidence of COVID-19 has increased markedly, making it difficult to meet the general time-in-range (TIR) requirement. Therefore, the investigators investigated a more clinically practical TIR threshold and examined its association with the prognosis of COVID-19 patients with type-2 diabetes.

participant population/health conditions：Participants were equipped with isCGM sensors on admission.

According to the outcome, the patients were divided into favorable outcome group and composite outcome group.

DETAILED DESCRIPTION:
patients with NCP who were discharged or died. Clinical data and blood glucose variability parameters were collected by computer blood glucose monitoring technology (CGM). Time in range (TIR), time above target range (TAR), time below target range (TBR), mean amplitude of glycemic excursions (MAGE), absolute mean daily difference (MODD) and other indicators were used.

ELIGIBILITY:
Inclusion Criteria:

1. All patients met the diagnostic criteria of type 2 diabetes mellitus in "Chinese Guidelines for the Prevention and treatment of type 2 Diabetes Mellitus (2020 edition)" formulated by the Chinese Diabetes Society of the Chinese Medical Association, and were previously diagnosed with type 2 diabetes mellitus and newly diagnosed with type 2 diabetes mellitus after admission
2. Patients with mild, moderate, severe and critical COVID-19 in accordance with the guidelines of "Diagnosis and Treatment of novel coronavirus Infection (Trial version 10)"
3. Patients receiving CGM or peripheral blood glucose monitoring during hospitalization

Exclusion Criteria:

1. Cases with incomplete data
2. Non-NCP and non-T2DM patients
3. Patients who did not receive CGM or peripheral blood glucose monitoring

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients with T2DM all had moderate or severe cases and were diagnosed according to the guidelines issued by the World Health Organization (WHO), meeting at least the following criteria: positive COVID-19 RNA PCR and characteristic imaging manifestations of novel coronavirus pneumonia.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
The composite adverse outcomes | Up to 3 weeks
  The composite adverse outcomes were defined as either a >20-day length of stay16 intensive care unit admission, mechanical ventilation use, or death.

CONTACTS AND LOCATIONS:
Overall Officials: Kuanxiao Tang, M.D., Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu hospital of shandong university, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided